CLINICAL TRIAL: NCT02049450
Title: A Single Arm, Multicenter, Phase IIa Study to Explore the Efficacy and Safety of Ruxolitinib (INC424) in Regularly Transfused Patients With Thalassemia
Brief Title: Study of Efficacy and Safety of INC424 in Regularly Transfused Patients With Thalassemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424X2201; 2013-002812-28 (EudraCT Number)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Thalassemia Major
Keywords: thalassemia; thalassemia major; spleen enlargement; INC424; ruxolitinib
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Splenomegaly | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INC424 (ruxolitinib) - Study Treatment (Experimental): Regularly transfused adult patients with thalassemia and spleen enlargement.
  Interventions: Drug: ruxolitinib

INTERVENTIONS:
Drug: ruxolitinib — Ruxolitinib was taken at a starting dose of 10 mg twice daily with dose adjustments within the range of 5 to 25 mg twice daily.
  Other Names: INC424

SUMMARY:
Patients with severe thalassemia (thalassemia major) present with severe anemia that required life-long transfusion therapy, spleen enlargement that led to increased transfusion requirement, and other serious complications as early death, growth retardation, bone deformations and iron overload due to blood transfusions. Splenectomy can significantly reduce transfusion requirement in thalassemia patients, but it is associated with an increased risk of serious complications such as sepsis and thrombosis. Preliminary preclinical and clinical data suggested that JAK2 inhibition, by reducing spleen size, could improve hemoglobin levels, thereby eliminating the need for splenectomy and reducing transfusion requirement and related iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thalassemia on a regular and stable transfusion regimen (at least 2 RBC units within every 4-week interval for 24 weeks prior to Screening) and anticipated to receive the same transfusion regimen during the study.
* Patients with spleen enlargement at Screening, defined as spleen palpable below the costal margin and spleen volume of ≥ 450 cm3 as confirmed by MRI (or CT scan in applicable patients).
* Patients need to be on iron chelation treatment (deferoxamine or deferasirox) for at least four weeks prior to Screening

Exclusion Criteria:

* Splenectomy prior to or planned during the study
* Active serious bacterial, mycobacterial, fungal, parasitic or viral infection which requires therapy (e.g., pneumonia, tuberculosis, systemic mycosis, herpes zoster)
* Hemoglobin <65 g/L (<4.0 mmol/L) at Screening
* Platelet count <75×109/L, absolute neutrophils count < 1.5×109/L at Screening.
* Estimated MDRD < 30 mL/min/1.73 m2 at Screening.
* ALT (SGPT) levels >5 times ULN at Screening.
* Hepatocellular disease such as hepatitis B (presence of HBs antigen), hepatitis C (presence of HCV RNA), liver cirrhosis.
* HIV positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, Athens, GR, Greece
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
- Novartis Investigative Site, Beirut, Lebanon
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 30 patients were planned to be enrolled in the study. 30 patients were analyzed in the full analysis, PK, and safety sets; 27 patients were analyzed in the per-protocol set.
Period: Overall Study
Arm/Group | INC424 (Ruxolitinib) - Study Treatment
Started | 30
Discontinued Treatment Prior to Week 30 | 4
Entered Extension Phase | 18 (Of 26 who completed Core phase 18 moved into Ext. phase; All 18 eventually discontinued Ext. phase)
Completed | 26 (Completed = Completed Core phase of study)
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Patients/guardian decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | INC424 (Ruxolitinib) - Study Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Change of Hematocrit Adjusted Volume of Red Blood Cells (RBC)
Description: Change of RBC transfusion requirement measured as percent change of the hematocrit-adjusted volume of transfused RBC and observed during within on-treatment interval (any time-points of RBC transfusion between week 6 and week 30 driven by the individual patient's need) compared to baseline (defined by pre-treatment interval between Week - 24 to start of treatment).
Time Frame: week 6 to week 30 interval
Population: Per-Protocol Set (PPS) consisted of a subset of patients in the Safety Set who were compliant with requirements of the Study Protocol. Patients were excluded from the PPS if: they had no or incomplete history of RBC transfusions within 24 weeks prior to the first dose of ruxolitinib or discontinued treatment with ruxolitinib prior to Week 18.
Measure: Mean (Standard Deviation); unit: % change of hematocrit-adjusted volume
Arm/Group | INC424 (Ruxolitinib) - Study Treatment
Number analyzed (Participants) | 27
% change of hematocrit-adjusted volume | -5.934 (22.1681)

2. Secondary Outcome: Percentage Change in Spleen Volume (cm3)
Description: Change of spleen volume from baseline at week 12 and week 30 as measured by magnetic imaging resonance (MRI) or computed tomography (CT).
Time Frame: baseline, week 12, week 30
Population: The Safety Set consisted of all patients who received at least one dose of ruxolitinib. All safety data was analyzed using the Safety set. The FAS and Safety set are identical in this study.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | INC424 (Ruxolitinib) - Study Treatment
Number analyzed (Participants) | 30
percentage change
  % change from baseline at Week 12: number analyzed (Participants) | 26
  % change from baseline at Week 12 | -19.733 (16.0539)
  % change from baseline at Week 30: number analyzed (Participants) | 25
  % change from baseline at Week 30 | -26.829 (16.6936)

3. Secondary Outcome: Percentage Change in Mean Pre-transfusion Hemoglobin by 6 Week Time Intervals
Description: Change from baseline in pre-transfusion hemoglobin levels
Time Frame: baseline, weeks 0 - 30
Population: The Safety Set consists of all patients who received at least one dose of ruxolitinib. All safety data was analyzed using the Safety set. The FAS and Safety set are identical in this study.
Measure: Mean (Standard Deviation); unit: percentage change of hemoglobin levels
Arm/Group | INC424 (Ruxolitinib) - Study Treatment
Number analyzed (Participants) | 30
percentage change of hemoglobin levels
  Weeks 0 - 6 ): number analyzed (Participants) | 27
  Weeks 0 - 6 ) | 0.43 (10.135)
  Weeks 6 - 12: number analyzed (Participants) | 27
  Weeks 6 - 12 | 2.87 (10.555)
  Weeks 12 - 18: number analyzed (Participants) | 27
  Weeks 12 - 18 | 2.78 (11.081)
  Weeks 18 - 24: number analyzed (Participants) | 26
  Weeks 18 - 24 | -0.56 (9.760)
  Weeks 24 - 30: number analyzed (Participants) | 26
  Weeks 24 - 30 | 0.06 (14.321)

4. Secondary Outcome: Percentage Change in Spleen Length (cm) Below the Left Coastal Margin
Description: Change of spleen length from baseline over time measured by palpitation by time
Time Frame: baseline, weeks 1,2,3,4,6,12,18,24,30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change in spleen length
Arm/Group | INC424 (Ruxolitinib) - Study Treatment
Number analyzed (Participants) | 30
percentage change in spleen length
  Week 1 | -11.19 (15.376)
  Week 2 | -22.11 (23.604)
  Week 3: number analyzed (Participants) | 29
  Week 3 | -25.01 (24.178)
  Week 4: number analyzed (Participants) | 29
  Week 4 | -26.94 (25.343)
  Week 6: number analyzed (Participants) | 29
  Week 6 | -33.85 (25.251)
  Week 12: number analyzed (Participants) | 29
  Week 12 | -49.29 (26.792)
  Week 18: number analyzed (Participants) | 27
  Week 18 | -56.32 (29.994)
  Week 24: number analyzed (Participants) | 27
  Week 24 | -56.93 (29.552)
  Week 30: number analyzed (Participants) | 24
  Week 30 | -57.40 (36.970)

5. Secondary Outcome: Pharmacokinetics (PK) Parameter of Cmin
Description: C min of INC424 by actual dose administered from 10mg bid to 20mg bid. Plasma PK samples were collected at Day 15 (Week 2), and Day 85 (Week 12). Cmin was collected immediately prior to dosing. n= number of patients with valid PK samples as per definition of the PK analysis set.
Time Frame: week 2, week 12
Population: The PK analysis set includes all patients with at least one evaluable PK sample at any visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 10 mg Bid: Patients who received INC422 10mg bid
- 15mg Bid: Patients who received INC422 15mg bid
- 20mg Bid: Patients who received INC422 20mg bid
Arm/Group | 10 mg Bid | 15mg Bid | 20mg Bid
Number analyzed (Participants) | 30 | 16 | 2
ng/mL
  Week 2 (Day 15): number analyzed (Participants) | 28 | 16 | 2
  Week 2 (Day 15) | 7.5800 (7.57959) | NA (NA) — N/A = per protocol, dose increase was not allowed prior to Week 6 so at week 2 no dose >10mg BID was expected | NA (NA) — N/A = per protocol, dose increase was not allowed prior to Week 6 so at week 2 no dose >10mg BID was expected
  Week 12 (Day 85): number analyzed (Participants) | 11 | 15 | 2
  Week 12 (Day 85) | 9.1300 (7.61039) | 18.5400 (23.99940) | 20.2300 (25.98617)

6. Secondary Outcome: Pharmacokinetics (PK) Parameter of Cmax
Description: Cmax (1h) of INC424 by actual dose administered from 10mg bid to 20mg bid. Plasma PK samples were collected at Day 1, Week 2, and Week 12. Cmax was collected within a +/- 1 hour post dose.
  n= number of patients with valid PK samples as per definition of the PK analysis set.
Time Frame: Day 1, Week 2 (Day 15), Week 12 (Day 85)
Population: The PK analysis set includes all patients with at least one evaluable PK sample at any visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 5mg Bid: Patients who received INC422 5mg bid
- 10mg Bid: Patients who received INC422 10mg bid
Arm/Group | 5mg Bid | 10mg Bid | 15mg Bid | 20mg Bid
Number analyzed (Participants) | 2 | 30 | 16 | 2
ng/mL
  Day 1: number analyzed (Participants) | 1 | 29 | 16 | 2
  Day 1 | 58.2000 (0.00) | 126.8000 (58.70337) | 0.00 (0.00) | 0.00 (0.00)
  Week 2: number analyzed (Participants) | 1 | 28 | 16 | 2
  Week 2 | 56.7000 (0.00) | 125.400 (40.61805) | 0.00 (0.00) | 0.00 (0.00)
  Week 12: number analyzed (Participants) | 2 | 11 | 16 | 2
  Week 12 | 0.00 (0.00) | 107.2100 (50.07525) | 245.6900 (50.00362) | 185.0000 (97.58074)

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Arm/Group | INC424 (Ruxolitinib) - Study Treatment
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INC424 (Ruxolitinib) - Study Treatment (N=30)
Anaemia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia viral (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INC424 (Ruxolitinib) - Study Treatment (N=30)
Anaemia (Blood and lymphatic system disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 3
Pyrexia (General disorders) | 2
Gastroenteritis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Weight increased (Investigations) | 5
Increased appetite (Metabolism and nutrition disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety